CLINICAL TRIAL: NCT05114486
Title: A Phase 3 Study of the Safety and Efficacy of 2% Pilocarpine Ophthalmic Spray Administered With the Optejet® Microdose Dispenser for Temporary Improvement of Near Vision in Adults With Presbyopia
Brief Title: Safety & Efficacy of Pilocarpine Ophthalmic Spray for Temporary Improvement of Near Vision in Presbyopic Adults
Acronym: VISION-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eyenovia Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: EYN-PRS-PI-32
Record Dates: First submitted 2021-11-05; First posted 2021-11-10 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pilocarpine 2% Ophthalmic Spray (Experimental): 2% pilocarpine ophthalmic spray administered with the Optejet dispenser
  Interventions: Combination Product: Pilocarpine Ophthalmic administered with the Optejet dispenser
- Placebo Spray (Placebo Comparator): Placebo ophthalmic spray administered with the Optejet dispenser
  Interventions: Combination Product: Placebo administered with the Optejet dispenser

INTERVENTIONS:
Combination Product: Pilocarpine Ophthalmic administered with the Optejet dispenser — Pilocarpine 2% ophthalmic spray administered with the Optejet dispenser
  Other Names: MicroLine
  Arms: Pilocarpine 2% Ophthalmic Spray
Combination Product: Placebo administered with the Optejet dispenser — Vehicle ophthalmic solution administered with the Optejet dispenser
  Arms: Placebo Spray

SUMMARY:
Volunteer participants are evaluated for eligibility during a Screening Visit; those meeting study inclusion/exclusion criteria are scheduled for 2 treatment visits. At each treatment visit, 1 of the 2 study treatments is self-administered to both eyes. Afterwards, efficacy and safety assessments are performed over a 3-hour period.

ELIGIBILITY:
Primary Inclusion Criteria:

* Poor near vision impacting daily living that requires near correction
* Best-corrected distance visual acuity (BCDVA) of 0.0 logMar or better
* Manifest refraction spherical equivalent ≥ -2.00 Diopters (D) and ≤ +2.00 D
* Monocular DCNVA between 0.4 and 0.7 logMAR, inclusive
* In need of near addition power < +2.00 D to achieve BCNVA of 0.0 logMAR

Primary Exclusion Criteria:

* Diagnosis of glaucoma or ocular hypertension
* Narrow iridocorneal angles
* History of intraocular surgery, refractive surgery, laser treatment, or iris surgery
* Clinically significant abnormality of cornea, lens, retina, ciliary body, or iris
* Presence/history of a severe/serious ocular condition or any other unstable medical condition
* Presence or history of manifest strabismus, amblyopia, or nystagmus
* Current active eye disease for which topical or systemic ophthalmic medication is necessary, except for dry eye syndrome managed using artificial tears
* Clinically significant external ocular inflammation within 30 days of Screening Visit
* Current use or history of rigid gas permeable (RGP) contact lens use within 30 days of Screening Visit
* Known pilocarpine allergy or contraindication to use of pilocarpine
* Presence or history of congenital heart anomaly, valve disease, or other cardiac disease
* Disabling arthritis or limited motor coordination that would limit the subject's ability to self-administer study solution using the Optejet

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects gaining ≥ 15 letters in mesopic, high contrast, binocular distance corrected near visual acuity (DCNVA) with ≤ 5 letter loss in mesopic, high contrast, binocular distance visual acuity (DVA) | 120 minutes post-dosing
  The proportion of subjects gaining ≥ 15 letters in mesopic, high contrast, binocular DCNVA with ≤ 5 letter loss DVA as compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Tsontcho (Sean) Ianchulev, MD, MPH, Study Chair — Eyenovia Inc.
Locations (9):
- United States (9):
  - VISION-2 Study Site #57, San Diego, California
  - VISION-2 Study Site #59, Fairfield, Connecticut
  - VISION-2 Study Site #56, Louisville, Kentucky
  - VISION-2 Study Site #19, Columbus, Ohio
  - VISION-2 Study Site #58, Philadelphia, Pennsylvania
  - VISION-2 Study Site #62, Sioux Falls, South Dakota
  - VISION-2 Study Site #55, Memphis, Tennessee
  - VISON-2 Study Site #60, Austin, Texas
  - VISION-2 Study Site #61, Draper, Utah

IPD SHARING:
Plan to Share IPD: No